CLINICAL TRIAL: NCT01817517
Title: Phase 1 Study of Thalamic Deep Brain Stimulation for the Treatment of Refractory Tourette Syndrome
Brief Title: Thalamic Deep Brain Stimulation for the Treatment of Refractory Tourette Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Expired in IRB
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00073086
Record Dates: First submitted 2013-03-18; First posted 2013-03-25 (Estimated); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deep Brain Stimulation implant (Experimental): Unblinded treatment arm, thalamic DBS for Tourette syndrome.
  Interventions: Device: Medtronic Activa Deep Brain Stimulation System

INTERVENTIONS:
Device: Medtronic Activa Deep Brain Stimulation System

SUMMARY:
This research is being performed to try to understand if the use of deep brain stimulation or DBS can treat the symptoms of Tourette syndrome that do not respond well to current medications. In order to do this the investigators will place small stimulation leads on both sides of the brain in a region (a portion of the thalamus) that may alter the abnormal activity in the brain contributing to the symptoms of Tourette syndrome. This requires two surgical procedures, and several preoperative and postoperative visits for tuning the stimulation parameters and recording stimulation effects. The FDA has not approved DBS for use in people with Tourette syndrome, and Medtronic (the manufacturer of the device) has not conducted testing for the system in Tourette syndrome. Therefore its use in this study is experimental.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females who are >=15 years of age. There is no strict age cutoff at the upper limit of inclusion, however subjects may meet the exclusion criteria based on medical contraindications to deep brain stimulation surgery (Points 3. and 6. under the Exclusion Criteria). For subjects in the age range of 15-24 years, an additional Ethics Committee consultation will be obtained prior to offering the subject the required screening visit. This is based on the revised screening criteria now proposed by Shrock, Mink, et al. on studies investigating DBS in TS. Additionally, for subjects in the age range of 15-20, a caregiver will be required to be present for all study visits.
2. Subject has a diagnosis of TS as determined by a review of medical records, discussion with referring psychiatrist as well as the DSM-IV criteria and videotaped assessment. This will include an assessment to determine the presence of psychogenic tics, embellishment, factitious symptoms, personality disorders and malingering.
3. Subject determined to be treatment-resistant for at least one year prior to the Screening Visit as demonstrated by clinical evidence (determined by review of medical records and discussion with referring psychiatrist or neurologist) of persistent functionally impairing tics that have not responded to treatment with a minimum of three adequate regimens of medication including two failed trials of at least one typical neuroleptic and one atypical neuroleptic medication, along with one failed trial of a first tier medication as defined as follows:

   1. Adequate trials of one non-neuroleptic medication including drugs from the following (first tier) list: clonidine, guanfacine, topiramate, baclofen, levetiracetam, and clonazepam. Trial failure is defined as demonstrated lack of efficacy or severe side effects.
   2. Two adequate trials of at least one typical neuroleptic medication (pimozide, fluphenazine, haloperidol) and at least one atypical neuroleptic (risperidone, aripiprazole, ziprasidone, olanzapine, quetiapine). Trial failure is defined as demonstrated lack of efficacy or severe side effects.
4. A mandatory trial of behavioral interventions in an attempt to reduce the severity of the tics or comorbid symptoms must also be completed by the subject before offering participation in this trial. This may include habit reversal therapies, stress reduction therapies, or other behavioral therapies under investigation for tic suppression.
5. Subject has both significant vocal and motor tics with a tic subscale score of at least 35 on the YGTSS (Yale Global Tic Severity Scale) at all three Baseline Visits prior to undergoing surgery. For subjects with predominantly vocal tics (and minimal motor) causing significant problems this score requirement will be reduced to 18, similarly for subjects with predominantly motor tics (and minimal vocal) causing significant problems the required score will be 18. A portion of the study team, including the surgeon and two neurologists, will determine by consensus which category the subject falls into and whether the tics are a significant problem.
6. All other aspects of the subject's care must be optimized during the preceding 6 months before admission to the study. This includes treatment for comorbid medical, neurological, and psychiatric disorders. Additionally, it includes psychological interventions for any ongoing psychosocial problems the subject may have during the preceding 6 months before study admission.
7. Subject must be ambulatory.
8. Females who are postmenopausal, physically incapable of childbearing, or practicing an acceptable method of birth control. Acceptable methods of birth control include surgical sterilization, hormonal contraceptives, or double-barrier methods (condom or diaphragm with a spermicidal agent or intrauterine device [IUD]). If practicing an acceptable method of birth control, a negative urine pregnancy test result has been obtained at baseline Visits 1 and 3.
9. Subject is determined by an independent psychiatrist with expertise in capacity assessments to have decision-making capacity to provide informed consent.
10. Subject is able to read English, understand and cooperate with study procedures, and has signed a written informed consent form prior to any study procedures.

Exclusion Criteria:

1. Subject has a positive urine drug screen at any of the three Baseline Visits.
2. Subject had major surgery within three months prior to Baseline Visit 1 or has other surgery planned during the proposed study period.
3. Subject is determined by medical consultant to have medical contraindications to undergoing surgery.
4. Subject is pregnant or breast-feeding.
5. Subject has a history of alcohol or drug abuse within the past 6 months and/or dependence within the past year.
6. Subject has a medical illness/condition, and/or abnormal diagnostic finding that would interfere with the completion of the study, confound the results of the study, or pose risk to the patient.
7. Subject has an untreated or uncontrolled Axis I disorder or other major psychiatric disorder including major depression, bipolar disorder, or schizophrenia as determined by the screening psychiatrist.
8. Subject has either a current or past history of suicidal plan and/or intent.
9. Subject has a tic disorder or other movement disorder attributable to another medical, neurological, or psychiatric disorder other than Tourette Syndrome.
10. Subject has a drug-induced tic disorder.
11. Subject has significant psychosocial factors that might increase the risk of the DBS procedure or complicate recovery and outcome assessments. (Examples include - history of noncompliance with previous medical and psychosocial treatments, multiple failed medication treatments of inadequate dose or duration, a history of multiple other surgical procedures with poor outcome, unexplained medical history gaps, or pending lawsuits or other legal action.)
12. Subject has metal in the head or any other type of implanted stimulator (i.e. cardiac pacemaker, deep brain stimulator for a different disease, spinal cord stimulator, cochlear implant, vagus nerve stimulator, etc.).
13. Subject has participated in another investigational drug trial or therapeutic trial within 30 days of Baseline Visit 1.
14. Subject has a diagnosis of intellectual disability with documented IQ<70.
15. Subject has a neurological condition, or a history of traumatic brain injury associated with loss of consciousness of > 1 hour and/or intracranial/epidural/subdural bleeding.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-03; Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ankur Butala, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Deep Brain Stimulation Implant: Unblinded treatment arm, thalamic DBS for Tourette syndrome.
  Medtronic Activa Deep Brain Stimulation System
Period: Overall Study
Arm/Group | Deep Brain Stimulation Implant
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Deep Brain Stimulation Implant
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2
Yale Global Tic Severity Scale (YGTSS) Total Score [Number; unit: units on a scale] — The Yale Global Tic Severity Scale (YGTSS) is clinician-administered used to assess severity of tics over the past week in individuals with Tourette Syndrome and other tic disorders. It evaluates motor and phonic tics across several dimensions-number, frequency, intensity, complexity, interference. Scores are combined to create Total Motor Tic score, Total Phonic Tic score, and combined Total Tic score, and separate Impairment scale providing a comprehensive measure of tic severity and impact on daily life. Total score range 0- 100. Higher score suggests worse severity of tics. Population: value for each subject is reported
  units on a scale
    Subject 1: number analyzed (Participants) | 1
    Subject 1 | 68
    Subject 2: number analyzed (Participants) | 1
    Subject 2 | 71
Yale Brown Obsessive Compulsive Score [Number; unit: units on a scale] — The Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) is a widely used clinical assessment tool for measuring the severity of obsessive-compulsive disorder (OCD) symptoms. The Y-BOCS consists of 10 items, 5 for obsessions and 5 for compulsions. Each item is rated on a 0-4 scale, with 0 indicating no symptoms and 4 indicating severe symptoms. A score range of 0-40. Higher is worse. Population: value for each subject is reported
  units on a scale
    Subject 1: number analyzed (Participants) | 1
    Subject 1 | 0
    Subject 2: number analyzed (Participants) | 1
    Subject 2 | 19
WHO Adult ADHD Self-Report Scale (ASRS) [Number; unit: units on a scale] — Total score range from 0 to 54. A higher score corresponds to a worse severity of ADHD Population: value for each subject is reported
  units on a scale
    Subject 1: number analyzed (Participants) | 1
    Subject 1 | 5
    Subject 2: number analyzed (Participants) | 1
    Subject 2 | 4
Grooved Pegboard Test - Dominant Hand [Number; unit: seconds] — The subject must place pegs shaped like keys into a board containing recesses that are oriented in randomly varying directions. The test is administered twice, once with the right and once with the left hand. Scores are time to completion in seconds for each hand and errors for each hand defined as number of pegs dropped during performance of the task. Lower scores (i.e. shorter duration in seconds) is preferred with normative data for age-matched controls. Population: value for each subject is reported
  seconds
    Subject 1: number analyzed (Participants) | 1
    Subject 1 | 80
    Subject 2: number analyzed (Participants) | 1
    Subject 2 | 58.5
Judgement of Line Orientation [Number; unit: score on a scale] — The Judgment of Line Orientation (JLO) test is a neuropsychological test that measures visuospatial skills, specifically the ability to judge and match the angles of lines. The test requires visually comparing and matching angled lines with an array of 11 choices. Two points are awarded for correctly identifying both target lines, for a total score range of 0-30 points. A higher score indicates better visuospatial ability, while a lower score suggests a deficit. Population: value for each subject is reported
  score on a scale
    Subject 1: number analyzed (Participants) | 1
    Subject 1 | 13
    Subject 2: number analyzed (Participants) | 1
    Subject 2 | 27
Time on Trail Making Test (TMT- A) [Number; unit: seconds] — The Time on Trails A (TMT) is scored by recording the number of seconds to complete each part of the test, with greater time indicating greater impairment. Normative ranges are used for interpretation and are stratified by age and education. TMT-A is an alphabetical sequence. A common benchmark for TMT-A is an average time of around 29 seconds, with a deficient score often considered to be over 78 seconds. Population: value for each subject is reported
  seconds
    Subject 1: number analyzed (Participants) | 1
    Subject 1 | 40
    Subject 2: number analyzed (Participants) | 1
    Subject 2 | 14
Time on Trail Making Test (TMT-B) [Number; unit: seconds] — The Time on Trails B (TMT) is scored by recording the number of seconds to complete each part of the test, with greater time indicating greater impairment. Normative ranges are used for interpretation and are stratified by age and education. TMT-B is an alternating alphabetical and numeral sequence. For TMT-B, the average is around 75 seconds, and a deficient score can be over 273 seconds. Population: value for each subject is reported
  seconds
    Subject 1: number analyzed (Participants) | 1
    Subject 1 | 480
    Subject 2: number analyzed (Participants) | 1
    Subject 2 | 25
Hopkins Verbal Learning Test - Delayed Free Recall [Number; unit: items recalled] — The Hopkins Verbal Learning Test-Revised (HVLT-R) is a brief, standardized neuropsychological test used to assess verbal memory and learning by having an individual recall and recognize a list of 12 words. It evaluates immediate recall, delayed recall, and delayed recognition over a 25-minute interval and is particularly useful for screening for memory problems. The total score range is 0 - 12, where 12 items were successfully and spontaneously recalled after 25 minutes. Population: value for each subject is reported
  items recalled
    Subject 1: number analyzed (Participants) | 1
    Subject 1 | 2
    Subject 2: number analyzed (Participants) | 1
    Subject 2 | 12
Verbal Fluency Test (COWAT) [Number; unit: total # of words (FAS)] — The Controlled Oral Word Association Test (COWAT) is a verbal fluency test that assesses spontaneous word production. The COWAT is scored by tallying the total number of acceptable generated within 60 seconds for three letters (e.g., F, A, S). The lowest possible score is zero, There is no limit to the higher end of the scale given that participants can produce as many words as possible for each of the three letters. Higher scores indicate greater word retrieval and better cognitive function Population: value for each subject is reported
  total # of words (FAS)
    Subject 1: number analyzed (Participants) | 1
    Subject 1 | 11
    Subject 2: number analyzed (Participants) | 1
    Subject 2 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Yale Global Tic Severity Scale (YGTSS)
Description: Investigators will assess deep brain stimulation effects on tic frequency and severity using the change in Yale Global Tic Severity Scale (YGTSS) in this population of Tourette syndrome patients. The scales range from 0-100, higher scores indicate greater tic severity and impairment.
Time Frame: 1 year after neurostimulator implantation
Population: values are per participant
Measure: Number; unit: Score on a scale
Arm/Group | Deep Brain Stimulation Implant
Number analyzed (Participants) | 2
Score on a scale
  Subject 1: number analyzed (Participants) | 1
  Subject 1 | 44
  Subject 2: number analyzed (Participants) | 1
  Subject 2 | 61

2. Primary Outcome: Number of Participants Free of Adverse Device Effects (ADEs).
Description: We will assess the incidence of adverse device effects (ADEs) as defined by the Code of Federal Regulations (21 CFR 812.3) at 1 year. Number of participants free of adverse events by 1year post implantation is reported.
Time Frame: 1 year after neurostimulator implantation.
Measure: Count of Participants; unit: Participants
Arm/Group | Deep Brain Stimulation Implant
Number analyzed (Participants) | 2
Participants | 2

3. Secondary Outcome: Change From Baseline in the Yale-Brown Obsessive Compulsive Scale
Description: We will assess deep brain stimulation effects on obsessive compulsive disorder symptoms using the Yale-Brown Obsessive Compulsive Scale (Baseline score - Final score). Score range 0-40, higher scores indicate greater severity of OCD symptoms.
Time Frame: 1 year after neurostimulator implantation.
Population: values are per participant
Measure: Number; unit: score on a scale
Arm/Group | Deep Brain Stimulation Implant
Number analyzed (Participants) | 2
score on a scale
  Subject 1: number analyzed (Participants) | 1
  Subject 1 | 0
  Subject 2: number analyzed (Participants) | 1
  Subject 2 | 5

4. Secondary Outcome: Change From Baseline in the WHO Adult ADHD Self-Report Scale (ASRS)
Description: We will assess deep brain stimulation effects on ADHD symptoms as measured by the WHO Adult ADHD Self-Report Scale (ASRS).
Time Frame: 1 year after neurostimulator implantation.
Population: values are per participant
Measure: Number; unit: score on a scale
Arm/Group | Deep Brain Stimulation Implant
Number analyzed (Participants) | 2
score on a scale
  Subject 1: number analyzed (Participants) | 1
  Subject 1 | 3
  Subject 2: number analyzed (Participants) | 1
  Subject 2 | -4

5. Other Pre Specified Outcome: Change From Baseline in the Grooved Pegboard Test
Description: We will assess deep brain stimulation effects on Grooved Pegboard test as a part of the neurocognitive assessment of this group of Tourette syndrome patients. We will measure change in seconds 1y after stimulation activation (of the dominant hand).
Time Frame: 1 year after neurostimulator implantation.
Population: Participants with data collected
Measure: Number; unit: seconds (reduction)
Arm/Group | Deep Brain Stimulation Implant
Number analyzed (Participants) | 1
seconds (reduction) | 4

6. Other Pre Specified Outcome: Change From Baseline in the Judgement of Line Orientation
Description: We will assess deep brain stimulation effects on the Judgement of Line Orientation test as a part of the neurocognitive assessment of this group of Tourette syndrome patients.
Time Frame: 1 year after neurostimulator implantation.
Measure: Number; unit: score on a scale
Arm/Group | Deep Brain Stimulation Implant
Number analyzed (Participants) | 1
score on a scale | 1

7. Other Pre Specified Outcome: Change From Baseline in the Trailmaking Test - A
Description: We will assess deep brain stimulation effects on the Trailmaking Test (A) as a part of the neurocognitive assessment of this group of Tourette syndrome patients.
Time Frame: 1 year after neurostimulator implantation.
Measure: Number; unit: seconds
Arm/Group | Deep Brain Stimulation Implant
Number analyzed (Participants) | 1
seconds | 10

8. Other Pre Specified Outcome: Change in Trail Making Test - B
Description: Change in seconds at 1 year on the Trail Making Test - Part B (Baseline score - Final Score). The Time on Trails B (TMT) is scored by recording the number of seconds to complete each part of the test, with greater time indicating greater impairment. Normative ranges are used for interpretation and are stratified by age and education. TMT-B is an alternating alphabetical and numeral sequence. For TMT-B, the average is around 75 seconds, and a deficient score can be over 273 seconds.
Time Frame: 1year
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change From Baseline in the Hopkins Verbal Learning Test
Description: We will assess deep brain stimulation effects on the change Hopkins Verbal Learning Test (delayed recall) as a part of the neurocognitive assessment of this group of Tourette syndrome patients. Note, a positive value indicates an improvement, a negative number worsening.
Time Frame: 1 year after neurostimulator implantation.
Measure: Number; unit: change # of items recalled
Arm/Group | Deep Brain Stimulation Implant
Number analyzed (Participants) | 1
change # of items recalled | -2

10. Other Pre Specified Outcome: Change From Baseline in the Verbal Fluency Test (COWAT)
Description: We will assess deep brain stimulation effects on the change of Verbal Fluency Test (COWAT) as a part of the neurocognitive assessment of this group of Tourette syndrome patients. Note, a positive value indicates an improvement, a negative number worsening.
Time Frame: 1 year after neurostimulator implantation.
Measure: Number; unit: change in total # of words (FAS)
Arm/Group | Deep Brain Stimulation Implant
Number analyzed (Participants) | 1
change in total # of words (FAS) | -6

ADVERSE EVENTS:
Time Frame: Immediately post implantation up to study termination (approximately 6 years 4 months)
Arm/Group | Deep Brain Stimulation Implant
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deep Brain Stimulation Implant (N=2)
Lead Fracture (Product Issues) | 1 (1) — DBS Electrode Fracture / Abnormal System Impedances
Meningoencephalitis (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study had recruitment limitations (both screened for consideration and implantations), partly due to staffing and administrative issues, which hampered analysis at a group level. Therefore, individual results were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT01817517/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT01817517/ICF_001.pdf